CLINICAL TRIAL: NCT06946134
Title: 18-Month Clinical Evaluation of Self-Adhesive Flowable Giomer Compared to Conventional Flowable Giomer in Carious Cervical Lesions: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amera Nabel, master holder, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CairoU PhD protocol for Amira
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cervical Caries
Keywords: Self-adhesive giomer; Bioactive; Randomized clinical trial.; USPHS criteria; Carious cervical lesion; Class V; Clinical performance; FIT SA; Beautifil Flow Plus
MeSH Terms: conditions — Root Caries | interventions — Beautifil Flow Plus F00

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beautifil Flow Plus F00 (Active Comparator): Conventional flowable giomer restorative material
  Interventions: Other: Beautifil Flow Plus F00
- FIT SA (Experimental): Self adhesive flowable giomer restorative material
  Interventions: Other: FIT SA

INTERVENTIONS:
Other: FIT SA — self-adhesive flowable giomer restorative material
  Arms: FIT SA
Other: Beautifil Flow Plus F00 — Conventional flowable giomer restorative material
  Arms: Beautifil Flow Plus F00

SUMMARY:
The material under investigation will offer the patient a high strength and high durability restoration with the advantage of having anti-bacterial properties.

DETAILED DESCRIPTION:
There is no available evidence for assessing FIT SA restorative material in restoration of cervical lesions. Therefore, this study aims to provide valuable insights into the shear bond strength and clinical performance, in terms of the biological, mechanical and esthetic parameters, of FIT SA restorative material in restoration of cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical carious lesions in anterior teeth and premolars
2. Small to moderate class V carious lesion (ICDAS 3 & 4).
3. Vital upper or lower periodontally sound teeth with no signs of irreversible pulpitis.
4. Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth

Exclusion Criteria:

1. Cervical carious lesions in molars.
2. Deep carious defects (close to pulp, less than 1 mm distance).
3. Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.
4. Non-vital teeth, Fractured or cracked teeth.
5. Endodontically treated teeth.
6. Periodontally affected teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance | 18 months
  Clinical Performance using Modified USPHS criteria

IPD SHARING:
Plan to Share IPD: Yes
There is no available evidence for assessing FIT SA restorative material in restoration of cervical lesions. Therefore, this study aims to provide valuable insights into the shear bond strength and clinical performance, in terms of the biological, mechanical and esthetic parameters, of FIT SA restorative material in restoration of cervical lesions

REFERENCES:
- See also: Related Info — https://doi.org/10.21608/EDJ.2024.267906.2924